CLINICAL TRIAL: NCT01986244
Title: Total Ankle Replacement for Ankle Arthritis
Acronym: TAR1600
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00001600
Record Dates: First submitted 2013-11-11; First posted 2013-11-18 (Estimated); Last update posted 2020-05-06 (Actual); Status verified 2020-05

CONDITIONS: Ankle Osteoarthritis
Keywords: Osteoarthritis; Arthritis; Joint Diseases
MeSH Terms: conditions — Osteoarthritis; Arthritis; Joint Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- STAR Total Ankle Replacement: Procedure: Total Ankle Replacement Surgery using the STAR
- Salto Talaris Total Ankle Replacement: Procedure: Total Ankle Replacement Surgery using the Salto Talaris
- In-Bone Total Ankle Replacement: Procedure: Total Ankle Replacement Surgery using the In-Bone

SUMMARY:
The purpose of this study is to prospectively evaluate the functional outcome and patient satisfaction of total ankle replacement for tibio-talar osteoarthritis.

DETAILED DESCRIPTION:
If a patient chooses to participate, they will be asked to sign the consent form and will be asked to complete the following patient outcome questionnaires: Visual Analog Pain Scale, Short-form 36, AOFAS hind foot score, and the Short Musculoskeletal Function Assessment questionnaire. The patient will then undergo surgery at a later date. Following surgery, the patient will present for routine follow-up appointments. At six month, one year, and yearly visits, the patients participating in the study will be asked to complete the previously mentioned outcome questionnaires. These are all normal follow-up visit time points; the patients will not be asked to return to clinic for any additional visits that would not be routine. At each visit, the patient will also receive plain x-rays. Plain x-rays are part of routine follow-up and not additional tests for this study. In addition, each patient will be tested pre-operatively as well as one year and two years post-operatively in order to gain a better understanding of the effect of total ankle replacements on lower extremity kinematics and kinetics. In order to understand the effect of the ankle replacement on lower extremity kinematics and kinetics, each subject will be asked to complete a series of functional tasks. First patients will be asked to complete a series of clinical tests to assess the patients ability to complete different balance tasks and walking trials. Patients will first be asked to stand with their legs approximately shoulder width apart on top of the one of the four force plates that are embedded in the ground in the lab. Patients will be asked to stand for at least 10 seconds. The time that they are able to remain balanced will be monitored as well as the movement of the center of pressure (COP) beneath the patient's feet. Each patient will then be asked to complete 3 other standing tasks on the force plate. These standing tasks will be a semi-tandem stance, tandem stance and single limb stance. The semi-tandem stance will require the patient to place one foot slightly in front of the other, but still side by side. The tandem stance will require the patients to place one foot in front of the other. Each of these tasks will be completed for 10 seconds or as long as possible while the COP is recorded. The second functional task to be completed is a four square step test. This test will consist of patients stepping forward, backward, and from side to side in order to assess their movement. This test will be timed from start to finish to see how long it takes for each patient to complete the task pre-operatively as well as post-operatively. Following the functional testing, each subject will have a series of reflective markers attached to different anatomical landmarks in order to monitor joint position and to be able to calculate joint moments during 3 different movement tasks. Once the markers have been placed patients will be asked to walk along a 10 meter walkway at a self selected speed which will be monitored using a timing system. In addition to a self-selected speed, each patient will be asked to walk at a standard speed of 1.3 m/s. Finally the patients will be asked to stand on both limbs and squat as far as possible as if sitting in a chair. Each of these tasks will be completed approximately seven times while lower extremity kinematics and kinetics will be recorded using an eight camera motion capture system and four force plates that are embedded within the 10 meter walkway. The only tests performed exclusively for research purposes will be the administered questionnaires and the gait analysis study. (The gait portion of this study is no longer being conducted.)

. The study will proceed until a minimum of 10-year follow-up is achieved for all patients. Questionnaires will be mailed out to the subjects at appropriate time points if they are unable to return to Duke.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (age > 18 years) who will benefit from a total ankle replacement, as determined by Drs. Nunley, DeOrio, Easley, or Adams, with the aid of the physical exam and routine radiography
* Treated at Duke University Medical Center
* Patients who have no medical conditions that would represent contraindications to surgery or anesthesia

Exclusion Criteria:

* Patients who do not meet the minimum age of 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients who will benefit from a total ankle replacement.
Sampling Method: Non-Probability Sample
Enrollment: 1043 (Actual)
Dates: Start 2007-06-13 (Actual); Primary Completion 2019-11-05 (Actual); Study Completion 2019-11-05 (Actual)

PRIMARY OUTCOMES:
Change in Visual Analog Pain Scale (VAS) | Preoperatively, 1yr, 2yr, 5yr, and 10yr
  To assess changes in pain across time following total ankle replacement across multiple time points. A visual analog scale of pain is an instrument used to measure the amount of pain a patient feels.
Change in Short Form Health Survey | Preoperatively, 1yr, 2yr, 5yr, and 10yr
  To assess functional health and well being across time following total ankle replacement and to determine if there are significant differences.
Change in Short Musculoskeletal Function Assessment (SMFA) | Preoperatively, 1yr, 2yr, 5yr, and 10yr
  SMFA is an outcome measure to provide a standardized measure of the actual physical limitations of the patient.
Change in AOFAS Hindfoot Scale questionnaire | Preoperatively, 1yr, 2yr, 5yr, and 10yr
  The AOFAS combines subjective scores of pain and function provided by the patient with objective scores based on the surgeon's physical examination of the patient.
Change in Foot and Ankle Disability Index (FADI) | Preoperatively, 1yr, 2yr, 5yr, and 10yr
  Patient reported function outcomes during activities of daily living.

SECONDARY OUTCOMES:
Changes in Three dimensional kinematic and kinetic assessments during level walking | preoperatively, 1yr, 2yr, 5yr, and 10yr
  In order to understand the effect of the ankle replacement on lower extremity kinematics and kinetics, each subject will be asked to complete a series of functional tasks and level walking trials at each of the study timepoints

CONTACTS AND LOCATIONS:
Overall Officials: James A Nunley, MD, Principal Investigator — Duke University
Locations (1):
- Duke Medical Plaza Page Road, Durham, North Carolina, United States